CLINICAL TRIAL: NCT05394402
Title: A Phase Ⅱ, Randomized, Double-blind, Placebo-controlled ， Evaluation of the Safety, Efficacy of SHR0410 Injection for Pain Management Following Orthopaedic Surgery
Brief Title: A Trial of SHR0410 Injection in Postsurgical Pain Management
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Adjustment of R&D strategy
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0410-202
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: SHR0410 Injection compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR0410 Injection High dose (Experimental)
  Interventions: Drug: SHR0410 Injection
- SHR0410 Injection Low dose (Experimental)
  Interventions: Drug: SHR0410 Injection
- Placebo for SHR0410 Injection (Placebo Comparator)
  Interventions: Drug: Placebo for SHR0410 Injection

INTERVENTIONS:
Drug: SHR0410 Injection — SHR0410 Injection
  Arms: SHR0410 Injection High dose; SHR0410 Injection Low dose
Drug: Placebo for SHR0410 Injection — SHR0410 Injection blank preparation
  Arms: Placebo for SHR0410 Injection

SUMMARY:
The study is being conducted to evaluate the efficacy, safety of SHR0410 Injection and to explore the reasonable of SHR0410 Injection for Pain Management after Orthopaedic Surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent；
2. Subjects requiring elective general anesthesia orthopedic surgery；
3. Male or female；
4. Meet the body mass index standard；
5. Conform to the ASA Physical Status Classification；
6. Negative pregnancy test.

Exclusion Criteria:

1. Subjects with a history of myocardial infarction or unstable angina pectoris；
2. Subjects with atrioventricular block or cardiac insufficiency；
3. Subjects with a history of malignancy ；
4. Subjects with a history of stroke；
5. Subjects with a history of mental illness；
6. Subjects with a history of difficult airway；
7. Random blood glucose ≥11.1mmol/L；
8. Subjects with poor blood pressure control；
9. Abnormal values in liver or renal function；
10. Subject with a history of substance abuse and drug abuse；
11. Allergic to drugs that may be used during the study；
12. Use other drugs that affect the analgesic effect before randomization, and the time from the last use to randomization is shorter than 5 half-lives；
13. Participated in clinical trials of other drugs (received experimental drugs)；
14. Other circumstances that the investigator judged inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Usage of Morphine, Post Surgery | 0 hour to 48 hours after IP administration
  Change in the amount of morphine use (in milligrams) by subjects in each treatment group for a 48 hour period post IP administration

SECONDARY OUTCOMES:
Usage of Morphine, Post Surgery at other intervals | 0 hour to 24 hours after IP administration ；24 hours to 48 hours after IP administration
  Change in the amount of morphine use (in milligrams) by subjects in each treatment group for 0-24 hours after IP administration.Change in the amount of morphine use (in milligrams) by subjects in each treatment group for 4-48 hours after IP administration.
the Sum of Pain Intensity Differences in Pain Score Over 6、12、24、48 、12-24、24-48 Hours under static condition | 48-hours
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Rating Scale (NRS), with higher numbers indicating a higher pain intensity, administered over 48 hours. Time weighted average change from baseline is calculated using the following: time weighted sum of pain intensity differences (SPID) divided by a constant (48 hours) to yield values on the 0-10 NRS.
the Sum of Pain Intensity Differences in Pain Score Over 6、12、24、48 、12-24、24-48 Hours under moving condition | 48-hours
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Rating Scale (NRS), with higher numbers indicating a higher pain intensity, administered over 48 hours. Time weighted average change from baseline is calculated using the following: time weighted sum of pain intensity differences (SPID) divided by a constant (48 hours) to yield values on the 0-10 NRS.
Time to First Dose of Rescue Analgesia | 0 hour to 48 hours after IP administration
  Time to first rescue was calculated as the elapsed time from administration of Dose 1 to the administration of the first dose of rescue analgesia.
Frequency of Doses of Rescue Analgesia Utilized Per Subject， total consumption of morphine Rescue Analgesia Utilized Per Subject | 0 hour to 24 hours after IP administration ；24 hours to 48 hours after IP administration ；0 hour to 48 hours after IP administration
  Rescue analgesia was available to subjects with inadequately controlled pain upon request.
Total press times of PCA pump and effective press times of PCA pump | 0 hour to 24 hours after IP administration ；24 hours to 48 hours after IP administration ；0 hour to 48 hours after IP administration
  Read and record the press times and effective press times from PCA
Proportion of subjects who did not receive Rescue Analgesia | 0 hour to 24 hours after IP administration ；24 hours to 48 hours after IP administration ；0 hour to 48 hours after IP administration
  Proportion of rescue was calculated as the elapsed time from administration of Dose 1 to the administration of the first dose of rescue analgesia.
Participant ' satisfaction score for analgesia treatment | 48-hours
  Participants recalled the postoperative analgesia effect and rated their satisfaction on a scale of 0 to 10, with 0 representing dissatisfied and 10 representing very satisfied.
Investigator satisfaction score for analgesia treatment | 48-hours
  Postoperative analgesia was evaluated by investigators. The scale ranges from 0 to 10, with 0 being dissatisfied and 10 being very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided